CLINICAL TRIAL: NCT06792019
Title: A Phase IB/II Clinical Study to Assess the Safety and Preliminary Efficacy of CM313(SC) Injection in Subjects With Platelet Transfusion Refractoriness
Brief Title: Study of CM313(SC) Injection in Subjects With Platelet Transfusion Refractoriness
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CM313-124102
Record Dates: First submitted 2025-01-15; First posted 2025-01-24 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Platelet Transfusion Refractoriness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CM313(SC)(low dose group) (Experimental)
  Interventions: Biological: CM313(SC) injection-low dose
- CM313(SC)(high dose group) (Experimental)
  Interventions: Biological: CM313(SC) injection-high dose

INTERVENTIONS:
Biological: CM313(SC) injection-low dose — Phase IB:CM313(SC) administered at low dose according to the protocol. Phase II:CM313(SC) administered at different doses based on Phase IB's results.
  Arms: CM313(SC)(low dose group)
Biological: CM313(SC) injection-high dose — Phase IB:CM313(SC) administered at high dose according to the protocol. Phase II:CM313(SC) administered at different doses based on Phase IB's results.
  Arms: CM313(SC)(high dose group)

SUMMARY:
This is a randomized, open-label, phase IB/II clinical study to evaluate the safety and preliminary efficacy of CM313(SC) injection in patients with Platelet Transfusion Refractoriness.

ELIGIBILITY:
Inclusion Criteria:

1. Thrombocytopenia dependent on platelet transfusions and diagnosed with platelet transfusion refractoriness.
2. Presence of one or more kinds of antiplatelet antibodies.
3. Male or female, age≥18 years.
4. The Eastern Cooperative Oncology Group (ECOG) physical status score ≤2.
5. Willing and able to comply with the requirements for this study and written informed consent.

Exclusion Criteria:

1. Diagnosed with Idiopathic thrombocytopenic purpura.
2. Platelet transfusion refractoriness caused by non-immune factors.
3. Previously treated with the anti-CD38 monoclonal antibody.
4. Have an allergy to humanized monoclonal antibody or any part of CM313.
5. Pregnant or breastfeeding females, or females planning to become pregnant during the study.
6. Any condition considered to be ineligible for the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2027-11-16 (Estimated); Study Completion 2027-11-16 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AE) | Up to 24 weeks
  Assess the safety of CM313(SC) injection

CONTACTS AND LOCATIONS:
Overall Officials: Jun Shi, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No